CLINICAL TRIAL: NCT02437890
Title: A Phase II Multicenter, Randomized, Double-blind, Placebo Controlled, Dose-range Finding Study to Evaluate the Safety and Efficacy of ALX-0061 Administered Subcutaneously in Subjects With Moderate to Severe Active Systemic Lupus Erythematosus
Brief Title: A Phase II Study to Evaluate Safety and Efficacy of ALX-0061 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0061-C204; 2015-000372-95 (EudraCT Number)
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — ALX-0061

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Two s.c. injections with placebo every 2 weeks (q2w).
  ***
  Placebo was supplied as a sterile liquid for s.c. injection at a volume of 0.5 mL and 1.0 mL in pre-filled single-use syringes. To maintain the blind, subjects randomly assigned to the placebo group received 2 s.c. injections q2w:
  Syringe A with placebo (1 mL) q2w starting at Day 1, up to and including Week 46.
  Syringe B with placebo (0.5 mL) q2w starting at Day 1, up to and including Week 46.
  Interventions: Biological: Placebo
- ALX-0061 75 mg q4w (Experimental): ALX-0061 75 mg every 4 weeks (q4w).
  ***
  Vobarilizumab (ALX-0061) and placebo were supplied as a sterile liquid for s.c. injection at a volume of 0.5 mL and 1.0 mL in pre-filled single-use syringes. To maintain the blind, subjects randomly assigned to ALX-0061 75 mg q4w received 2 s.c. injections q2w:
  Syringe A with placebo (1 mL) q2w starting at Day 1, up to and including Week 46.
  Syringe B with ALX-0061 (0.5 mL) q4w at Day 1, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44, and syringe B with placebo (0.5 mL) q4w at Weeks 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42, and 46.
  Interventions: Biological: ALX-0061; Biological: Placebo
- ALX-0061 150 mg q4w (Experimental): ALX-0061 150 mg every 4 weeks (q4w).
  ***
  Vobarilizumab (ALX-0061) and placebo were supplied as a sterile liquid for s.c. injection at a volume of 0.5 mL and 1.0 mL in pre-filled single-use syringes. To maintain the blind, subjects randomly assigned to ALX-0061 150 mg q4w received 2 s.c. injections q2w:
  Syringe A with ALX-0061 (1 mL) q4w at Day 1, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44, and syringe A with placebo (1 mL) q4w at Weeks 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42, and 46.
  Syringe B with placebo (0.5 mL) q2w starting at Day 1, up to and including Week 46.
  Interventions: Biological: ALX-0061; Biological: Placebo
- ALX-0061 150 mg q2w (Experimental): ALX-0061 150 mg every 2 weeks (q2w).
  ***
  Vobarilizumab (ALX-0061) and placebo were supplied as a sterile liquid for s.c. injection at a volume of 0.5 mL and 1.0 mL in pre-filled single-use syringes. To maintain the blind, subjects randomly assigned to ALX-0061 150 mg q2w received 2 s.c. injections q2w:
  Syringe A with ALX-0061 (1 mL) q2w starting at Day 1, up to and including Week 46.
  Syringe B with placebo (0.5 mL) q2w starting at Day 1, up to and including Week 46.
  Interventions: Biological: ALX-0061; Biological: Placebo
- ALX-0061 225 mg q2w (Experimental): ALX-0061 225 mg every 2 weeks (q2w).
  ***
  Vobarilizumab (ALX-0061) was supplied as a sterile liquid for s.c. injection at a volume of 0.5 mL and 1.0 mL in pre-filled single-use syringes. To maintain the blind, subjects randomly assigned to ALX-0061 225 mg q2w received 2 s.c. injections q2w:
  Syringe A with ALX-0061 (1 mL) q2w starting at Day 1, up to and including Week 46.
  Syringe B with ALX-0061 (0.5 mL) q2w starting at Day 1, up to and including Week 46.
  Interventions: Biological: ALX-0061

INTERVENTIONS:
Biological: ALX-0061
  Arms: ALX-0061 150 mg q2w; ALX-0061 150 mg q4w; ALX-0061 225 mg q2w; ALX-0061 75 mg q4w
Biological: Placebo
  Arms: ALX-0061 150 mg q2w; ALX-0061 150 mg q4w; ALX-0061 75 mg q4w; Placebo

SUMMARY:
Primary objective:

To assess the efficacy and safety of different dose regimens of ALX-0061 administered subcutaneously (s.c.) to subjects with moderate to severe active, seropositive systemic lupus erythematosus (SLE) compared to placebo.

Secondary objectives:

To assess the pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, flare rate, steroid reduction and health-related quality of life, with different dose regimens of ALX-0061.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman ≥ 18 years and < 65 years of age
2. Have a diagnosis of SLE for at least 6 months prior to screening and fulfill the 1997 American College of Rheumatology (ACR) or 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria
3. Have moderate to severe active SLE
4. Have seropositive disease at screening
5. Subject must be at least on one or more of the treatments for SLE as listed in the protocol
6. Others as defined in the protocol

Exclusion Criteria:

1. Have an A score on the revised BILAG-2004 other than in the mucocutaneous and/or musculoskeletal system at screening and at baseline for the organ systems that can be clinically assessed
2. Have a systemic inflammatory disease other than SLE
3. Clinically significant infection treated or needing treatment
4. Any active or recurrent viral infection that based on the Investigator´s clinical assessment makes the subject unsuitable for the study
5. Have received prior therapy blocking the interleukin-6 (IL-6) pathway
6. Others as defined in the protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Ablynx NV
Locations (117):
- United States (27):
  - Investigator Site, Birmingham, Alabama
  - Investigator Site, Glendale, Arizona
  - Investigator Site, Phoenix, Arizona
  - Investigator Site, Tucson, Arizona
  - Investigator Site, Artesia, California
  - Investigator Site, La Jolla, California
  - Investigator Site, La Palma, California
  - Investigator Site, Los Angeles, California
  - Investigator Site, Upland, California
  - Investigator Site, Aventura, Florida
  - Investigator Site, Clearwater, Florida
  - Investigator Site, Orlando, Florida
  - Investigator Site, Pinellas Park, Florida
  - Investigator Site, Atlanta, Georgia
  - Investigator Site, Stockbridge, Georgia
  - Investigator Site, Louisville, Kentucky
  - Investigator Site, Cumberland, Maryland
  - Investigator Site, Lansing, Michigan
  - Investigator Site, New York, New York
  - Investigator Site, Smithtown, New York
  - Investigator Site, Syracuse, New York
  - Investigator Site, Charlotte, North Carolina
  - Investigator Site, Raleigh, North Carolina
  - Investigator Site, Pittsburgh, Pennsylvania
  - Investigator Site, Jackson, Tennessee
  - Investigator Site, Austin, Texas
  - Investigator Site, Houston, Texas
- Argentina (6):
  - Investigator Site, Caba, Buenos Aires
  - Investigator Site, Caba
  - Investigator Site, Ciudad Autónoma de Buenos Aire
  - Investigator Site, Córdoba
  - Investigator Site, San Juan
  - Investigator Site, San Miguel de Tucumán
- Chile (2):
  - Investigator Site 1, Santiago
  - Investigator Site 2, Santiago
- Investigator Site, Prague, Czechia
- Germany (4):
  - Investigator Site, Berlin
  - Investigator Site, Dresden
  - Investigator Site, Mainz
  - Investigator Site, Mannheim
- Hungary (5):
  - Investigator Site 1, Budapest
  - Investigator Site 2, Budapest
  - Investigator Site, Debrecen
  - Investigator Site, Gyula
  - Investigator Site, Zalaegerszeg
- Mexico (7):
  - Investigator Site 1, Guadalajara
  - Investigator Site 2, Guadalajara
  - Investigator Site 3, Guadalajara
  - Investigator Site, Mexicali
  - Investigator Site, Mexico City
  - Investigator Site, Mérida
  - Investigator Site, San Luis Potosí City
- Peru (4):
  - Investigator Site 1, Lima
  - Investigator Site 2, Lima
  - Investigator Site 3, Lima
  - Investigator Site 4, Lima
- Philippines (6):
  - Investigator Site 1, Cebu City
  - Investigator Site 2, Cebu City
  - Investigator Site, Lipa City
  - Investigator Site, Makati City
  - Investigator Site, Manila
  - Investigator Site, Quezon City
- Poland (7):
  - Investigator Site, Bydgoszcz
  - Investigator Site, Katowice
  - Investigator Site 1, Lodz
  - Investigator Site 2, Lodz
  - Investigator Site 1, Poznan
  - Investigator Site 2, Poznan
  - Investigator Site, Szczecin
- Portugal (5):
  - Investigator Site, Almada
  - Investigator Site, Amadora
  - Investigator Site, Lisbon
  - Investigator Site, Ponte de Lima
  - Investigator Site, Porto
- Russia (9):
  - Investigator Site, Kazan'
  - Investigator Site, Kemerovo
  - Investigator Site, Orenburg
  - Investigator Site, Ryazan
  - Investigator Site 1, Saint Petersburg
  - Investigator Site 2, Saint Petersburg
  - Investigator Site, Smolensk
  - Investigator Site, Vladimir
  - Investigator Site, Voronezh
- Serbia (6):
  - Investigator Site 1, Belgrade
  - Investigator Site 2, Belgrade
  - Investigator Site 3, Belgrade
  - Investigator Site 4, Belgrade
  - Investigator Site 5, Belgrade
  - Investigator Site, Niška Banja
- South Korea (4):
  - Investigator Site, Daegu
  - Investigator Site, Gwangju
  - Investigator Site 1, Seoul
  - Investigator Site 2, Seoul
- Spain (8):
  - Investigator Site, A Coruña
  - Investigator Site 1, Barcelona
  - Investigator Site 2, Barcelona
  - Investigator Site 3, Barcelona
  - Investigator Site, Bilbao
  - Investigator Site 1, Madrid
  - Investigator Site 2, Madrid
  - Investigator Site, Sant Joan Despí
- Taiwan (5):
  - Investigator Site, Kaohsiung City
  - Investigator Site 1, Taichung
  - Investigator Site 2, Taichung
  - Investigator Site, Taipei
  - Investigator Site, Taoyuan District
- Ukraine (11):
  - Investigator Site, Ivano-Frankivsk
  - Investigator Site, Kharkiv
  - Investigator Site, Kryvyi Rih
  - Investigator Site 1, Kyiv
  - Investigator Site 2, Kyiv
  - Investigator Site 3, Kyiv
  - Investigator Site, Lviv
  - Investigator Site 1, Poltava
  - Investigator Site 2, Poltava
  - Investigator Site 1, Vinnytsia
  - Investigator Site 2, Vinnytsia

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 312 subjects were randomized at 91 sites located in Europe (37 sites; 155 subjects), Asia-Pacific (19 sites, 53 subjects), North America (21 sites; 52 subjects), and Latin America (14 sites, 52 subjects). Consent was obtained from the first subject on 02 July 2015; the last subject completed the final visit on 25 January 2018.
Pre-assignment Details: Of the 568 subjects screened, 256 were screen failures and 312 were randomly assigned to treatment (modified Intent-to-treat [mITT] population). All subjects received study drug and were included in the safety population. Overall, 254 subjects were included in the Per Protocol (PP) population.
Period: Overall Study
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Started | 62 | 64 | 62 | 62 | 62
Completed | 54 | 48 | 47 | 40 | 46
Not Completed | 8 | 16 | 15 | 22 | 16
Not completed — Non-compliance to study drug | 0 | 1 | 0 | 0 | 1
Not completed — Sponsor's decision | 1 | 1 | 4 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Unable to attend visit(s) | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 0 | 3 | 1
Not completed — Adverse Event | 4 | 9 | 5 | 11 | 7
Not completed — Withdrawal by Subject | 1 | 2 | 6 | 5 | 5
Not completed — Death | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Two s.c. injections with placebo every 2 weeks (q2w)
- ALX-0061 75 mg q4w: ALX-0061 75 mg every 4 weeks (q4w)
- ALX-0061 150 mg q4w: ALX-0061 150 mg every 4 weeks (q4w)
- ALX-0061 150 mg q2w: ALX-0061 150 mg every two weeks (q2w)
- ALX-0061 225 mg q2w: ALX-0061 225 mg every two weeks (q2w)
- Total: Total of all reporting groups
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | Total
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 64 | 62 | 62 | 62 | 312
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.11) | 42.0 (11.00) | 41.8 (10.79) | 39.2 (11.58) | 42.0 (10.44) | 41.4 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 61 | 61 | 57 | 300
  Male | 2 | 3 | 1 | 1 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 17 | 11 | 13 | 66
  Not Hispanic or Latino | 49 | 52 | 45 | 51 | 49 | 246
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 4 | 4 | 3 | 3 | 4 | 18
  Hungary | 2 | 4 | 2 | 2 | 4 | 14
  United States | 10 | 11 | 10 | 11 | 10 | 52
  Czechia | 2 | 1 | 0 | 0 | 3 | 6
  Philippines | 1 | 3 | 4 | 3 | 2 | 13
  Ukraine | 5 | 6 | 7 | 8 | 7 | 33
  Portugal | 2 | 2 | 0 | 1 | 1 | 6
  Russia | 3 | 6 | 5 | 8 | 6 | 28
  Spain | 3 | 2 | 2 | 1 | 0 | 8
  South Korea | 1 | 1 | 0 | 2 | 1 | 5
  Taiwan | 3 | 1 | 1 | 0 | 2 | 7
  Poland | 4 | 5 | 3 | 6 | 5 | 23
  Mexico | 5 | 6 | 5 | 5 | 5 | 26
  Chile | 0 | 1 | 1 | 0 | 0 | 2
  Serbia | 14 | 11 | 17 | 11 | 10 | 63
  Peru | 2 | 0 | 2 | 1 | 1 | 6
  Germany | 1 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects Who Achieved a Response at Week 24 According to the Modified British Isles Lupus Assessment Group (BILAG)-Based Composite Lupus Assessment (mBICLA) Score
Description: The primary endpoint was evaluated by determining if there was a dose-response relationship between the mBICLA response rate at Week 24 and the dose administered, using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. The existence of several candidate parametric models was assumed and multiple comparison techniques were used to choose the model(s) most likely to represent the true underlying dose-response curve. The selected model could further be used to guide the choice of adequate doses.
  mBICLA responders were defined as subjects who met all of the following criteria:
  1. BILAG-2004 normal improvement: all A scores at Baseline improved to B, C or D, and all B scores improved to C or D.
  2. No worsening in disease activity: no new BILAG-2004 A scores and ≤ 1 new increase to B.
  3. No worsening of total mSLEDAI-2K score from Baseline.
  4. No significant deterioration (< 10% worsening from Baseline) in PGA.
  5. No treatment failure (including the premature
Time Frame: At Week 24 visit
Population: mITT Population - Non-response imputation (NRI)
Measure: Count of Participants; unit: Participants
Groups:
- ALX-0061 150 mg q2w: ALX-0061 150 mg every 2 weeks (q2w)
- ALX-0061 225 mg q2w: ALX-0061 225 mg every 2 weeks (q2w)
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants | 29 | 28 | 24 | 24 | 23
Statistical Analysis 1: Comparison: Placebo vs ALX-0061 75 mg q4w vs ALX-0061 150 mg q4w vs ALX-0061 150 mg q2w vs ALX-0061 225 mg q2w; A multiple contrast test was used to establish evidence of a drug effect by testing for a statistically significant dose-response signal for clinical endpoint and patient population investigated in the study. Candidate dose-response models were selected amongst the following types of parametric models: linear model, Emax model, logistic model, a 1st Beta model, and a 2nd Beta model. Model tested: linear model; Test type: Superiority; p = 0.526, Multiple Contrast Test — Threshold for statistical significance: p = 0.05
Statistical Analysis 2: Comparison: Placebo vs ALX-0061 75 mg q4w vs ALX-0061 150 mg q4w vs ALX-0061 150 mg q2w vs ALX-0061 225 mg q2w; A multiple contrast test was used to establish evidence of a drug effect by testing for a statistically significant dose-response signal for clinical endpoint and patient population investigated in the study. Candidate dose-response models were selected amongst the following types of parametric models: linear model, Emax model, logistic model, a 1st Beta model, and a 2nd Beta model. Model tested: Emax model; Test type: Superiority; p = 0.504, Multiple Contrast Test — Threshold for statistical significance: p = 0.05
Statistical Analysis 3: Comparison: Placebo vs ALX-0061 75 mg q4w vs ALX-0061 150 mg q4w vs ALX-0061 150 mg q2w vs ALX-0061 225 mg q2w; A multiple contrast test was used to establish evidence of a drug effect by testing for a statistically significant dose-response signal for clinical endpoint and patient population investigated in the study. Candidate dose-response models were selected amongst the following types of parametric models: linear model, Emax model, logistic model, a 1st Beta model, and a 2nd Beta model. Model tested: logistic model; Test type: Superiority; p = 0.548, Multiple Contrast Test — Threshold for statistical significance: p = 0.05
Statistical Analysis 4: Comparison: Placebo vs ALX-0061 75 mg q4w vs ALX-0061 150 mg q4w vs ALX-0061 150 mg q2w vs ALX-0061 225 mg q2w; A multiple contrast test was used to establish evidence of a drug effect by testing for a statistically significant dose-response signal for clinical endpoint and patient population investigated in the study. Candidate dose-response models were selected amongst the following types of parametric models: linear model, Emax model, logistic model, a 1st Beta model, and a 2nd Beta model. Model tested: 1st Beta model; Test type: Superiority; p = 0.985, Multiple Contrast Test — Threshold for statistical significance: p = 0.05
Statistical Analysis 5: Comparison: Placebo vs ALX-0061 75 mg q4w vs ALX-0061 150 mg q4w vs ALX-0061 150 mg q2w vs ALX-0061 225 mg q2w; A multiple contrast test was used to establish evidence of a drug effect by testing for a statistically significant dose-response signal for clinical endpoint and patient population investigated in the study. Candidate dose-response models were selected amongst the following types of parametric models: linear model, Emax model, logistic model, a 1st Beta model, and a 2nd Beta model. Model tested: 2nd Beta model; Test type: Superiority; p = 0.524, Multiple Contrast Test — Threshold for statistical significance: p = 0.05

2. Secondary Outcome: Number and Percentage of Subjects With mBICLA Response at Week 24 and Week 48
Description: Number and percentage of mBICLA responders at Week 24 and Week 48
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 61 | 64 | 58 | 62 | 61
  Week 24 | 28 | 28 | 22 | 24 | 22
  Week 48: number analyzed (Participants) | 59 | 61 | 60 | 60 | 60
  Week 48 | 28 | 32 | 22 | 19 | 22

3. Secondary Outcome: Number and Percentage of Subjects With Modified Systemic Lupus Erythematosus Responder Index (mSRI-4) Response at Week 24 and Week 48
Description: The composite index mSRI-4 enables quantification of decrease and increase in disease activity in a broad spectrum of manifestations thereby offering a comprehensive assessment of SLE disease status. mSRI combines advantages from 3 validated measurement tools. The mSRI-4 criteria for response are:
  1. modified SLE disease activity index 2000 (mSLEDAI-2K): ≥ 4 point reduction (covers global disease improvement),
  2. British Isles Lupus Assessment Group 2004 (BILAG-2004): no new A domain score and no more than 1 new increase to B (covers organ-specific disease improvement),
  3. Physician's Global Assessment (PGA) (is used as validity and safety net for items that were not addressed by the other two indices): < 10% increase from Baseline (no worsening) When all 3 criteria are met, the subject is a mSRI-4 responder at that time point.
  Subjects who were treatment failures or discontinued from treatment were considered non-responder after treatment failure/discontinuation.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 59 | 63 | 58 | 61 | 60
  Week 24 | 37 | 39 | 30 | 33 | 29
  Week 48: number analyzed (Participants) | 58 | 60 | 59 | 58 | 60
  Week 48 | 34 | 36 | 29 | 26 | 33

4. Secondary Outcome: Number and Percentage of Subjects With mSRI-5 Response at Week 24 and Week 48
Description: The mSRI-5 criteria for response are:
  1. mSLEDAI-2K: ≥ 5 point reduction
  2. BILAG-2004: no new A domain score and no more than 1 new increase to B domain score
  3. PGA: no worsening (< 10% increase from Baseline) Only subjects with Baseline mSLEDAI-2K ≥ 5 were considered for the derivation of that endpoint.
  Subjects who were treatment failures or discontinued from treatment were considered non-responder after treatment failure/discontinuation.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 57 | 61 | 54 | 59 | 58
  Week 24 | 17 | 24 | 19 | 20 | 16
  Week 48: number analyzed (Participants) | 56 | 58 | 55 | 56 | 58
  Week 48 | 20 | 28 | 18 | 16 | 22

5. Secondary Outcome: Number and Percentage of Subjects With mSRI-6 Response at Week 24 and Week 48
Description: The mSRI-6 criteria for response are:
  1. mSLEDAI-2K: ≥ 6 point reduction
  2. BILAG-2004: no new A domain score and no more than 1 new increase to B domain score
  3. PGA: no worsening (< 10% increase from Baseline) Only subjects with Baseline mSLEDAI-2K ≥ 6 were considered for the derivation of that endpoint.
  Subjects who were treatment failures or discontinued from treatment were considered non-responder after treatment failure/discontinuation
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 57 | 61 | 54 | 59 | 58
  Week 24 | 16 | 23 | 19 | 19 | 15
  Week 48: number analyzed (Participants) | 56 | 58 | 55 | 56 | 58
  Week 48 | 20 | 28 | 16 | 16 | 22

6. Secondary Outcome: Number and Percentage of Subjects With mSRI-7 Response at Week 24 and Week 48
Description: The mSRI-7 criteria for response are:
  1. mSLEDAI-2K: ≥ 7 point reduction
  2. BILAG-2004: no new A domain score and no more than 1 new increase to B domain score
  3. PGA: no worsening (< 10% increase from Baseline) Only subjects with Baseline mSLEDAI-2K ≥ 7 were considered for the derivation of that endpoint.
  Subjects who were treatment failures or discontinued from treatment were considered non-responder after treatment failure/discontinuation.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 46 | 47 | 39 | 50 | 43
  Week 24 | 9 | 8 | 8 | 12 | 7
  Week 48: number analyzed (Participants) | 46 | 45 | 40 | 47 | 42
  Week 48 | 12 | 14 | 7 | 8 | 9

7. Secondary Outcome: Number and Percentage of Subjects With mSRI-8 Response at Week 24 and Week 48.
Description: The mSRI-8 criteria for response are:
  1. mSLEDAI-2K: ≥ 8 point reduction
  2. BILAG-2004: no new A domain score and no more than 1 new increase to B domain score
  3. PGA: no worsening (< 10% increase from Baseline) Only subjects with Baseline mSLEDAI-2K ≥ 8 were considered for the derivation of that endpoint.
  Subjects who were treatment failures or discontinued from treatment were considered non-responder after treatment failure/discontinuation.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 45 | 47 | 37 | 49 | 42
  Week 24 | 9 | 7 | 8 | 10 | 7
  Week 48: number analyzed (Participants) | 45 | 45 | 38 | 46 | 41
  Week 48 | 11 | 14 | 7 | 7 | 8

8. Secondary Outcome: Change From Baseline in Modified Systemic Lupus Erythematosus Disease Activity Index 2000 (mSLEDAI-2K) Score at Week 24 and Week 48
Description: The Systemic Lupus Erythematosus Disease Activity Index 2000 is a 1-page weighted score for 24 items (seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, hematuria, proteinuria, pyuria, rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, etc). The manifestations felt to be most commonly contributing to disease activity are included and scored based on the presence (= 1 multiplied by weight) or absence (= 0) within 30 days prior to the evaluation. The total score ranges from 0-105 (= sum of individual scores), with 105 being higher disease activity. mSLEDAI-2K derives from the standard index by omitting low complement. Mean changes from baseline were derived from an ANCOVA model with treatment as factor and baseline mSLEDAI-2K Score and geographic region as covariates. A negative change from baseline reflects an improvement.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 24: number analyzed (Participants) | 53 | 50 | 51 | 48 | 51
  Week 24 | -4.0 (0.42) | -4.6 (0.43) | -3.8 (0.43) | -4.3 (0.44) | -3.6 (0.44)
  Week 48: number analyzed (Participants) | 51 | 46 | 47 | 36 | 45
  Week 48 | -4.5 (0.40) | -5.2 (0.43) | -4.3 (0.42) | -4.9 (0.48) | -4.9 (0.44)

9. Secondary Outcome: Number and Percentage of Subjects With BILAG-2004 Normal Improvement at Week 24 and Week 48
Description: Normal Improvement: all A scores at baseline improved to B/C/D, and all B scores improved to C or D.
  Only subjects with non-missing BILAG-2004 who had at least one A or B score at Baseline were assessed for this endpoint
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | 31 | 29 | 28 | 25 | 24
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 34 | 34 | 29 | 22 | 25

10. Secondary Outcome: Number and Percentage of Subjects With BILAG-2004 Enhanced Improvement at Week 24 and Week 48
Description: Enhanced improvement: all A scores at baseline improved to B/C/D, and all B scores improved to C or D and no worsening between consecutive visits from baseline up to the considered visit Only subjects with non-missing BILAG-2004 who had at least one A or B score at Baseline were assessed for this endpoint
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | 7 | 16 | 11 | 6 | 13
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 45
  Week 48 | 5 | 10 | 7 | 6 | 7

11. Secondary Outcome: BILAG-2004 Total Score at Baseline, Week 24 and Week 48
Description: The British Isles Lupus Assessment Group 2004 (BILAG-2004) is a comprehensive composite clinical index that has been developed based on the principle of a physician's intention to treat using a nominal consensus approach. In the index, the nine systems (not organs) considered are: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, renal, ophthalmic and hematological. Disease activity in each of the nine systems is categorized into five levels: grades A (= severe disease activity requiring systemic high dose oral corticosteroids, i.v. pulse corticosteroids, etc.) to E (= system never involved).
  BILAG total score is derived by assigning the following value to each grade and summing the sores over all organ systems:
  A = 12, B = 8, C = 1, D/E = 0. The total score ranges from 0-108, with 108 representing high disease activity in all 9 systems requiring high doses of corticosteroids, starting/increasing immunosuppressive drugs, etc.
Time Frame: At Baseline, Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Baseline | 17.4 (0.78) | 17.9 (0.69) | 15.2 (0.68) | 17.4 (0.71) | 17.3 (0.82)
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | 6.8 (0.78) | 5.7 (0.79) | 7.0 (0.76) | 7.2 (0.94) | 7.4 (0.84)
  Week 48: number analyzed (Participants) | 53 | 48 | 50 | 39 | 45
  Week 48 | 6.0 (0.73) | 4.0 (0.72) | 5.2 (0.74) | 6.0 (0.92) | 6.2 (0.91)

12. Secondary Outcome: Number and Percentage of Subjects With BILAG-2004 Normal Improvement in Mucocutaneous System at Week 24 and Week 48
Description: An improvement is defined as an A score at Baseline improved to B/C/D, or a B score improved to C or D.
  Only subjects with non-missing BILAG-2004 who had at least one A or B score at Baseline were assessed for this endpoint
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 47 | 45 | 43 | 43 | 47
  Week 24 | 25 | 24 | 18 | 21 | 25
  Week 48: number analyzed (Participants) | 45 | 41 | 37 | 34 | 40
  Week 48 | 26 | 27 | 18 | 18 | 22

13. Secondary Outcome: Number and Percentage of Subjects With BILAG-2004 Normal Improvement in Musculoskeletal System at Week 24 and Week 48
Description: as for outcome 12
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 47 | 44 | 43 | 45 | 45
  Week 24 | 41 | 39 | 36 | 36 | 33
  Week 48: number analyzed (Participants) | 45 | 40 | 40 | 37 | 38
  Week 48 | 40 | 38 | 35 | 33 | 31

14. Secondary Outcome: Number and Percentage of Subjects With Persistent Minimal or no Activity in 9 Organ Systems According to BILAG-2004 Systems Tally at Week 24 and Week 48
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | 15 | 24 | 19 | 16 | 16
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 20 | 27 | 23 | 16 | 19

15. Secondary Outcome: Change From Baseline in Physician's Global Assessment (PGA) at Week 24 and Week 48
Description: The physician makes a mark between 0 ("no disease") and 100 mm ("severe disease") on the visual analogue scale (VAS) to indicate disease activity (independent of the subject's self-assessment).
  Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline PGA score and geographic region as covariates.
  A negative change from baseline reflects an improvement.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score on a scale
  Week 24: number analyzed (Participants) | 56 | 52 | 55 | 49 | 54
  Week 24 | -25.2 (2.03) | -28.4 (2.09) | -26.2 (2.04) | -23.5 (2.16) | -22.7 (2.08)
  Week 48: number analyzed (Participants) | 54 | 48 | 48 | 39 | 46
  Week 48 | -28.3 (1.73) | -32.9 (1.82) | -30.2 (1.82) | -30.1 (2.00) | -30.5 (1.87)

16. Secondary Outcome: Change From Baseline in Patient's Global Assessment at Week 24 and Week 48
Description: The subject makes a mark between 0 ("very good") and 100 mm ("very bad") on the VAS to indicate how the subject is doing, while considering all the ways SLE affects him/her.
  Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline Patient's Global Assessment and geographic region as covariates.
  A negative change from baseline reflects an improvement.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score on a scale
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 53
  Week 24 | -12.4 (2.87) | -13.5 (2.96) | -14.9 (2.87) | -20.1 (3.05) | -16.0 (2.98)
  Week 48: number analyzed (Participants) | 54 | 48 | 49 | 39 | 46
  Week 48 | -15.1 (2.70) | -21.5 (2.87) | -22.1 (2.82) | -27.2 (3.12) | -25.9 (2.94)

17. Secondary Outcome: Change From Baseline in Proteinuria at Week 24 and Week 48
Description: Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline proteinuria and geographic region as covariates
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: g/mol
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
g/mol
  Week 24: number analyzed (Participants) | 48 | 44 | 48 | 42 | 42
  Week 24 | 6.17 (3.730) | 1.77 (3.847) | 1.03 (3.735) | -3.02 (3.876) | 0.16 (3.962)
  Week 48: number analyzed (Participants) | 43 | 37 | 42 | 30 | 36
  Week 48 | 4.89 (5.732) | 3.83 (6.152) | -1.62 (5.761) | -0.49 (6.582) | -1.21 (6.191)

18. Secondary Outcome: Number of Subjects Who Were Treatment-emergent Urine Sediment Positive at Week 24 and Week 48
Description: Efficacy Laboratory Parameters (Urinalysis) - Active Urine Sediment Number of subjects who were urine sediment negative at Baseline, but positive at Week 24 and Week 48, respectively.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | 1 | 0 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 24 and Week 48
Description: Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline serum creatinine and geographic region as covariates
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
umol/L
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 53
  Week 24 | -1.25 (2.172) | -3.29 (2.237) | -1.50 (2.182) | -3.98 (2.309) | -0.86 (2.276)
  Week 48: number analyzed (Participants) | 54 | 47 | 50 | 38 | 46
  Week 48 | 1.19 (2.016) | -1.87 (2.152) | -6.26 (2.085) | -4.04 (2.359) | -1.24 (2.199)

20. Secondary Outcome: Change From Baseline in Creatinine Clearance Estimation (eGFR) at Week 24 and Week 48
Description: Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline eGFR and geographic region as covariates
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: mL/min/1.73m2
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
mL/min/1.73m2
  Week 24: number analyzed (Participants) | 55 | 52 | 56 | 49 | 53
  Week 24 | -1.63 (2.869) | 4.83 (2.931) | -1.72 (2.854) | -0.90 (3.044) | -8.91 (3.014)
  Week 48: number analyzed (Participants) | 53 | 47 | 50 | 38 | 46
  Week 48 | -6.00 (3.052) | 2.47 (3.231) | 4.66 (3.125) | -1.47 (3.562) | -8.08 (3.326)

21. Secondary Outcome: Number of and Percentage Treatment Failures From Baseline to Week 24 and Week 48
Description: Defined as non-protocol allowed increase in steroid dose, start i.v. or i.m. steroids, or start or increase of immunosuppressant
Time Frame: From Baseline to Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Baseline to Week 24 | 2 | 0 | 4 | 2 | 3
  Baseline to Week 48 | 5 | 1 | 9 | 6 | 6

22. Secondary Outcome: Number and Percentage of Subjects Experiencing Severe Flares According to BILAG-2004 Flare Index From Baseline to Week 24 and Week 48
Time Frame: From Baseline to Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Baseline to Week 24 | 8 | 6 | 6 | 7 | 6
  Baseline to Week 48 | 8 | 6 | 10 | 9 | 9

23. Secondary Outcome: Number and Percentage of Subjects Experiencing Severe Flares According to mSLEDAI-2K Flare Index (mSFI) From Baseline to Week 24 and Week 48
Time Frame: From Baseline to Week 24 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  Baseline to Week 24 | 1 | 0 | 2 | 2 | 1
  Baseline to Week 48 | 4 | 0 | 4 | 4 | 2

24. Secondary Outcome: Percent Change From Baseline in Daily Dose of Steroids at Week 24 and Week 48
Description: Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline prednisone equivalent total daily dose and geographic region as covariates
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
percentage
  Week 24: number analyzed (Participants) | 48 | 43 | 51 | 43 | 48
  Week 24 | 3.87 (2.781) | -0.80 (2.922) | 0.25 (2.689) | -1.40 (2.940) | -3.46 (2.831)
  Week 48: number analyzed (Participants) | 46 | 40 | 45 | 34 | 40
  Week 48 | 6.93 (5.047) | -3.22 (5.397) | -1.03 (5.050) | -2.32 (5.758) | -1.73 (5.521)

25. Secondary Outcome: Number and Percentage of Subjects Whose Daily Dose of Steroids Was Reduced Without Severe Flares During Weeks 40-48
Description: Number and percentage of subjects whose prednisone equivalent dose was >7.5 mg/day at baseline and reduced to ≤7.5 mg/day during Weeks 40-48 without experiencing a BILAG-2004-defined or mSFI-defined severe flare after the first prednisone equivalent dose decrease.
Time Frame: Between Week 40 and Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  BILAG-2004-defined Flare: number analyzed (Participants) | 34 | 36 | 30 | 32 | 36
  BILAG-2004-defined Flare | 3 | 2 | 5 | 1 | 3
  mSFI-defined Flare: number analyzed (Participants) | 34 | 36 | 30 | 32 | 36
  mSFI-defined Flare | 3 | 2 | 4 | 1 | 4

26. Secondary Outcome: Number and Percentage of Subjects Who Discontinued Prednisone (or Equivalent) by Week 48 Without Experiencing a Severe Flare
Description: Number and percentage of subjects who discontinued Prednisone (or equivalent) by Week 48 without experiencing a BILAG-2004-defined or mSFI-defined severe flare
Time Frame: Up to and including Week 48
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants
  BILAG-2004-defined Flare: number analyzed (Participants) | 54 | 52 | 55 | 54 | 56
  BILAG-2004-defined Flare | 0 | 0 | 1 | 1 | 0
  mSFI-defined Flare: number analyzed (Participants) | 54 | 52 | 55 | 54 | 56
  mSFI-defined Flare | 0 | 0 | 2 | 1 | 0

27. Secondary Outcome: Change From Baseline in Physical Component Scores of Short Form (36) Health Survey (SF-36) at Week 24 and Week 48
Description: The Short Form (36) Health Survey (SF-36) consists of 36 items that can be summarized into 8 domains: physical functioning, role limitations due to physical health problems (role-physical), bodily pain, general health, vitality, social functioning, role limitations due to emotional problems (role-emotional), and mental health. Two summary measures, the physical component summary and the mental component summary, can be derived based on these domain scores. Each score is directly transformed into a 0-100 score on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
  Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline SF-36 Score and geographic region as covariates. A positive change denotes an improvement.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 53
  Week 24 | 4.71 (1.241) | 4.56 (1.286) | 6.77 (1.242) | 4.67 (1.321) | 5.01 (1.292)
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 3.73 (1.414) | 6.97 (1.510) | 8.67 (1.460) | 8.62 (1.633) | 8.85 (1.535)

28. Secondary Outcome: Change From Baseline in Mental Component Scores of SF-36 at Week 24 and Week 48
Description: as for outcome 27
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 53
  Week 24 | 0.08 (0.703) | -0.99 (0.724) | -0.56 (0.703) | 0.45 (0.749) | -1.18 (0.732)
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 1.50 (0.716) | -0.58 (0.756) | -0.07 (0.737) | -1.07 (0.827) | -2.02 (0.777)

29. Secondary Outcome: Change From Baseline in 28 Joint Count Swollenness (SJC28) Score at Week 24 and Week 48
Description: Twenty-eight joints are assessed for swollenness (a score of 1 for a joint denotes a presence of swollenness). The sum is derived to create a total score (ranging from 0 to 28; where the highest score indicate all 28 joints are swollen). Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline SJC28 Score and geographic region as covariates. A negative change denotes an improvement.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | -4.8 (0.31) | -5.0 (0.32) | -4.9 (0.31) | -4.8 (0.33) | -4.5 (0.32)
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | -5.0 (0.28) | -5.4 (0.30) | -4.7 (0.29) | -5.1 (0.32) | -4.5 (0.30)

30. Secondary Outcome: Change From Baseline in 28 Joint Count Tenderness (TJC28) Score at Week 24 and Week 48
Description: Twenty-eight joints are assessed for tenderness (a score of 1 for a joint denotes a presence of tenderness). The sum is derived to create a total score (ranging from 0 to 28; where the highest score indicate all 28 joints are tender). Mean changes from baseline were derived from an analysis of covariance (ANCOVA) model with treatment as factor and baseline TJC28 Score and geographic region as covariates. A negative change denotes and improvement.
Time Frame: At Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 54
  Week 24 | -6.8 (0.49) | -6.8 (0.50) | -6.4 (0.49) | -5.8 (0.52) | -5.5 (0.50)
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | -6.6 (0.43) | -7.4 (0.46) | -6.4 (0.45) | -6.6 (0.50) | -6.5 (0.47)

31. Secondary Outcome: Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score at Week 12, Week 24 and Week 48
Description: CLASI Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and nonscarring alopecia. Evaluation of erythema and scale/hyperkeratosis is based on a table: rows represent anatomical areas and columns represent major clinical symptoms. The extent of involvement for each of the skin symptoms is documented for each anatomic area (erythema: 0=absent, 1=pink, 2=red, 3=dark red; scale: 0=absent, 1=scale, 2=verrucous/hypertrophic). Mucous membrane involvement and acute hair loss are scored based on the presence (=1) or absence (=0).
  Nonscarring alopecia is scored as 0=absent, 1=diffuse/non-inflammatory, 2=focal or patchy in 1 quadrant, 3=focal or patchy in >1 quadrant. The total score ranges from 0-70, with higher scores indicating more severe skin disease.
  Mean changes from baseline were derived from an ANCOVA model with treatment as factor and baseline CLASI Activity Score and geographic region as covariates. Negative change = improvement
Time Frame: At Week 12, Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 12: number analyzed (Participants) | 26 | 25 | 18 | 21 | 24
  Week 12 | -2.4 (0.53) | -1.9 (0.57) | -1.4 (0.65) | -1.6 (0.63) | -1.3 (0.57)
  Week 24: number analyzed (Participants) | 25 | 21 | 17 | 19 | 23
  Week 24 | -1.1 (0.53) | -2.1 (0.60) | -1.6 (0.66) | -1.3 (0.65) | -1.8 (0.57)
  Week 48: number analyzed (Participants) | 24 | 18 | 16 | 14 | 21
  Week 48 | -1.3 (0.59) | -3.0 (0.70) | -2.5 (0.73) | -2.1 (0.80) | -3.0 (0.64)

32. Secondary Outcome: Change From Baseline in CLASI Damage Score at Week 12, Week 24 and Week 48
Description: CLASI Damage is scored based on dyspigmentation and scarring. Evaluation of dyspigmentation and scarring is based on a table: rows represent anatomical areas and columns represent major clinical symptoms. The extent of involvement for each of the skin symptoms is documented for each anatomic area (dyspigmentation: 0=absent, 1=present; scarring: 0=absent, 1=scarring, 2=severely atrophic scarring or panniculitis). Subjects are also asked whether dyspigmentation due to SLE lesions usually remains visible for >12 months, which is considered permanent and results in doubling of the dyspigmentation score. Scarring alopecia is scored as follows: 0=absent, 3=1 quadrant, 4=2 quadrants, 5=3 quadrants, 6=affects the whole skull. Total score ranges from 0-56, with higher scores indicating more damaged skin.
  Mean changes from baseline were derived from an ANCOVA model with treatment as factor and baseline CLASI Damage Score and geographic region as covariates. Negative change = improvement.
Time Frame: At Week 12, Week 24 and Week 48
Population: mITT Population
Measure: Mean (Standard Error); unit: score
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
score
  Week 12: number analyzed (Participants) | 11 | 14 | 8 | 13 | 13
  Week 12 | 0.1 (0.49) | 0.1 (0.47) | -0.1 (0.59) | -0.3 (0.52) | -0.4 (0.52)
  Week 24: number analyzed (Participants) | 11 | 11 | 8 | 11 | 12
  Week 24 | 0.4 (0.61) | -0.4 (0.61) | -0.4 (0.73) | 0.3 (0.67) | -0.1 (0.66)
  Week 48: number analyzed (Participants) | 11 | 9 | 8 | 8 | 11
  Week 48 | 0.0 (0.57) | -0.1 (0.60) | -0.3 (0.68) | 0.4 (0.68) | -0.7 (0.63)

33. Secondary Outcome: ALX-0061 Serum Concentrations at Week 24 and Week 48
Time Frame: At Week 24 and Week 48
Population: Safety Population
Measure: Geometric Mean (Standard Deviation); unit: µg/mL
Groups:
- ALX-0061 75 mg 4qw: ALX-0061 75 mg every 4 weeks (q4w)
Arm/Group | ALX-0061 75 mg 4qw | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 64 | 62 | 62 | 62
µg/mL
  Week 24: number analyzed (Participants) | 43 | 53 | 47 | 50
  Week 24 | 0.118 (2.29) | 2.05 (3.89) | 18.1 (1.60) | 30.7 (1.62)
  Week 48: number analyzed (Participants) | 33 | 43 | 32 | 42
  Week 48 | 0.155 (3.28) | 2.17 (3.45) | 17.9 (1.71) | 36.1 (1.46)

34. Secondary Outcome: Actual Values of Soluble Interleukin 6 Receptor (sIL-6R) Concentrations at Baseline, Week 24, and Week 48
Time Frame: At Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
ng/mL
  Baseline: number analyzed (Participants) | 62 | 63 | 62 | 62 | 60
  Baseline | 42.22 (2.496) | 37.63 (1.933) | 38.10 (1.895) | 42.14 (3.366) | 36.92 (1.810)
  Week 24: number analyzed (Participants) | 55 | 51 | 54 | 49 | 53
  Week 24 | 39.70 (1.934) | 198.26 (18.856) | 603.51 (31.678) | 668.57 (25.568) | 634.49 (23.638)
  Week 48: number analyzed (Participants) | 53 | 47 | 50 | 38 | 46
  Week 48 | 39.41 (2.270) | 224.66 (25.515) | 610.86 (29.445) | 650.73 (38.516) | 659.79 (32.862)

35. Secondary Outcome: Actual Values of C-reactive Protein (CRP) Concentrations at Baseline, Week 24, and Week 48
Time Frame: At Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
nmol/L
  Baseline | 43.58 (9.527) | 49.05 (12.924) | 38.89 (8.394) | 66.32 (17.221) | 32.23 (4.957)
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 53
  Week 24 | 59.43 (11.277) | 47.22 (9.607) | 26.08 (9.995) | 3.83 (0.668) | 3.20 (0.357)
  Week 48: number analyzed (Participants) | 54 | 46 | 50 | 38 | 46
  Week 48 | 30.70 (4.709) | 37.65 (8.647) | 23.20 (6.705) | 4.41 (0.988) | 4.02 (0.962)

36. Secondary Outcome: Actual Values of Fibrinogen Concentrations at Baseline, Week 24, and Week 48
Time Frame: At Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
g/L
  Baseline | 3.2 (0.09) | 3.2 (0.08) | 3.2 (0.09) | 3.2 (0.10) | 3.1 (0.09)
  Week 24: number analyzed (Participants) | 55 | 52 | 54 | 49 | 51
  Week 24 | 3.3 (0.08) | 3.3 (0.10) | 2.3 (0.12) | 1.9 (0.05) | 1.9 (0.05)
  Week 48: number analyzed (Participants) | 51 | 48 | 49 | 36 | 46
  Week 48 | 3.3 (0.09) | 3.3 (0.12) | 2.3 (0.11) | 1.9 (0.06) | 1.9 (0.05)

37. Secondary Outcome: Actual Values of Anti-double-stranded (ds) DNA Concentrations at Baseline, Week 24, and Week 48
Time Frame: at Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
IU/mL
  Baseline | 132.90 (54.467) | 145.87 (113.907) | 52.88 (17.283) | 68.92 (23.226) | 73.34 (25.940)
  Week 24: number analyzed (Participants) | 55 | 52 | 55 | 49 | 53
  Week 24 | 81.36 (30.376) | 68.27 (35.053) | 46.99 (33.534) | 14.98 (4.499) | 23.25 (6.417)
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 81.80 (24.143) | 59.48 (32.190) | 74.21 (48.030) | 9.13 (2.108) | 15.53 (6.069)

38. Secondary Outcome: Actual Values of Complement C3 Concentrations at Baseline, Week 24, and Week 48
Time Frame: At Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
mg/dL
  Baseline | 102.3 (3.82) | 100.2 (4.12) | 101.9 (3.79) | 105.8 (4.38) | 98.6 (3.98)
  Week 24: number analyzed (Participants) | 55 | 52 | 55 | 47 | 52
  Week 24 | 101.7 (4.30) | 95.7 (3.81) | 82.0 (3.68) | 75.3 (2.90) | 71.8 (2.82)
  Week 48: number analyzed (Participants) | 53 | 48 | 50 | 38 | 45
  Week 48 | 95.8 (4.25) | 93.2 (4.20) | 79.0 (3.25) | 83.2 (3.18) | 72.3 (2.61)

39. Secondary Outcome: Actual Values of Complement C4 Concentrations at Baseline, Week 24, and Week 48
Time Frame: At Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
mg/dL
  Baseline | 17.3 (1.08) | 17.8 (1.07) | 15.9 (0.96) | 18.7 (1.19) | 16.3 (1.04)
  Week 24: number analyzed (Participants) | 54 | 52 | 55 | 47 | 52
  Week 24 | 17.5 (1.09) | 17.4 (1.10) | 10.6 (0.85) | 8.7 (0.40) | 7.9 (0.37)
  Week 48: number analyzed (Participants) | 52 | 47 | 48 | 38 | 43
  Week 48 | 16.3 (1.15) | 17.3 (1.27) | 10.5 (0.84) | 9.8 (0.89) | 8.1 (0.41)

40. Secondary Outcome: Actual Values for Hemolytic Complement Component 50 (CH50) at Baseline, Week 24, and Week 48
Time Frame: At Baseline, Week 24, and Week 48
Population: Safety Population
Measure: Mean (Standard Error); unit: unit(s)
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
unit(s)
  Baseline | 101.1 (7.46) | 109.6 (8.83) | 98.9 (6.95) | 103.0 (7.47) | 82.4 (7.09)
  Week 24: number analyzed (Participants) | 56 | 52 | 56 | 49 | 53
  Week 24 | 95.8 (7.94) | 107.0 (7.08) | 73.6 (6.94) | 56.7 (4.91) | 41.1 (3.63)
  Week 48: number analyzed (Participants) | 54 | 48 | 50 | 39 | 46
  Week 48 | 102.2 (8.38) | 113.1 (8.63) | 73.5 (8.26) | 68.4 (6.95) | 41.9 (3.32)

41. Secondary Outcome: Number and Percentage of Subjects Who Were Treatment-emergent (TE) Anti-drug Antibody (ADA) Positive
Time Frame: From first administration of ALX-0061 up to and including follow-up
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 62 | 64 | 62 | 62 | 62
Participants | 32 | 16 | 18 | 31 | 38

ADVERSE EVENTS:
Time Frame: From time of first study drug administration until the subject's study completion/discontinuation date.
Arm/Group | Placebo | ALX-0061 75 mg q4w | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64 | 0/62 | 2/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 7/62 | 2/64 | 4/62 | 5/62 | 5/62
Other Adverse Events (participants affected / at risk) | 40/62 | 40/64 | 31/62 | 47/62 | 44/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=62) | ALX-0061 75 mg q4w (N=64) | ALX-0061 150 mg q4w (N=62) | ALX-0061 150 mg q2w (N=62) | ALX-0061 225 mg q2w (N=62)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculoma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=62) | ALX-0061 75 mg q4w (N=64) | ALX-0061 150 mg q4w (N=62) | ALX-0061 150 mg q2w (N=62) | ALX-0061 225 mg q2w (N=62)
Urinary tract infection (Infections and infestations) | 8 (11) | 5 (10) | 7 (10) | 3 (5) | 8 (12)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (7) | 5 (5) | 5 (8) | 3 (5)
Nasopharyngitis (Infections and infestations) | 6 (8) | 6 (7) | 5 (6) | 2 (3) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3) | 2 (3) | 4 (4) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 3 (6) | 0 (0) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (3) | 2 (5) | 5 (17) | 5 (11)
Injection site rash (General disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (17) | 3 (6)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (16) | 4 (27) | 3 (4) | 3 (6) | 10 (10)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (6) | 3 (3) | 5 (9) | 6 (7)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 3 (4) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, in particular point 30, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-05-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT02437890/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT02437890/SAP_003.pdf